CLINICAL TRIAL: NCT02543164
Title: Comparison of the Glycemic Response of Consumption of Bread Enriched With Barley Beta-glucans With White Bread. Controlled Intervention Trial. A Pilot Study
Brief Title: Influence of Beta-glucan Enriched Barley Flour in Bread on Glycemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: Valens Int. d.o.o., Slovenija (Industry)
Responsible Party: Principal Investigator, Snežana Kocijančič, Ms., Institute of Nutrition, Slovenia (Nutris)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: KME68/02/15
Record Dates: First submitted 2015-09-01; First posted 2015-09-07 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Glycemic Index
Keywords: Glycemic Index; glycemic response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- REFERENCE: white bread (Other): Participants will consume a meal standardised to contain 50 g of available carbohydrates. Sample Will be consumed together with 250 mL of water, within 10-15 minutes.
  Interventions: Other: REFERENCE: white bread
- TEST: b-glucan enriched bread (Other): Participants will consume a meal standardised to contain 50 g of available carbohydrates. Sample Will be consumed together with 250 mL of water, within 10-15 minutes.
  Interventions: Other: TEST: b-glucan enriched bread

INTERVENTIONS:
Other: REFERENCE: white bread — Determination of glycemic response after consumption of white bread:
  Capillary glucose will be taken at 0 min (baseline sample), followed by 15, 30, 45, 60, 90 and 120 min after starting to eat the meal to calculate the area under the curve (AUC).
  Arms: REFERENCE: white bread
Other: TEST: b-glucan enriched bread — Determination of glycemic response after consumption of bread enriched with barley beta-glucans (Test A) :
  Capillary glucose will be taken at 0 min (baseline sample), followed by 15, 30, 45, 60, 90 and 120 min after starting to eat the meal to calculate the area under the curve (AUC).
  Arms: TEST: b-glucan enriched bread

SUMMARY:
Objective of the study is to investigate the influence of beta-glucan enriched barley flour as constituent of bread on glycaemic response (GR) in healthy human volunteers. Glycaemic response will be measured as AUC of blood glucose after consumption of barley bread, and compared with white bread.

DETAILED DESCRIPTION:
Objective of the study is to investigate the influence of beta-glucan enriched barley flour as constituent of bread on glycaemic response (GR) in healthy human volunteers. Glycaemic response will be measured as the area under the curve (AUC) of blood glucose after consumption of barley bread(s), and compared with AUC for white bread. Measurements will be done in line with recommendations. In line with recommendations ten healthy human volunteers will be tested to obtain a sufficient statistical power. GR measurement will be based on available carbohydrates. Amount of bread will be standardised to contain 50 g of available carbohydrates. Subjects will consume bread sample with 250 mL of water, within 10-15 minutes. Blood sampling times will be at 0 min (baseline sample), followed by 15, 30, 45, 60, 90 and 120 min after starting to eat the test meal. Glucose levels will be measured in capillary blood. For reference and test meals, the investigators will do at least 2 AUC measurements per subject. AUC calculation will be based on incremental AUC, ignoring area under the baseline. Comparison will be done as the mean of the individual ratios.

The differences between the different products ingested will be analyzed with the statistical test of analysis of variance. In case of failure to find homogeneity in the variances the nonparametric ANOVA, the Kruskal-Wallis test, will be used. The results will be expressed as mean ± standard deviation for each with a significance level of 0.05 for all the statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Willingness' to participate, self-diagnosed as healthy
* Age: 18-65 years

Exclusion Criteria:

* Allergy or intolerances to ingredients of tested products (bread)
* Renal impairment
* Diagnosed diabetes
* Level of glucose above 5.6mmol/l at first measurement
* Thyroid disease
* Use of medicines for lowering blood fats and/or preparations for weight loss or reducing the absorption of nutrients from the digestive tract

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Reduced area under the curve (AUC) of blood glucose levels in bread enriched with barley beta-glucans (reduced glycemic response) | up to 60 days (1 day experiments)
  Glycaemic response will be measured as the area under the curve (AUC) of blood glucose after consumption of barley bread(s), and compared with AUC for white bread. Blood sampling times will be at 0 min (baseline sample), followed by 15, 30, 45, 60, 75, 90 and 120 min after starting to eat the test meal. Glucose levels will be measured in capillary blood. AUC calculation will be based on incremental AUC, ignoring area under the baseline. Comparison will be done as the mean of the individual ratios. Primary outcome measure is significant reducment of AUC for bread enriched with barley beta-glucans (P<0.05).

CONTACTS AND LOCATIONS:
Overall Officials: Igor Pravst, Study Chair — Institute of Nutrition, Slovenia (Nutris); Snežana Kocijančič, Principal Investigator — Institute of Nutrition, Slovenia (Nutris)

REFERENCES:
- [Background] Brouns F, Bjorck I, Frayn KN, Gibbs AL, Lang V, Slama G, Wolever TM. Glycaemic index methodology. Nutr Res Rev. 2005 Jun;18(1):145-71. doi: 10.1079/NRR2005100. PMID 19079901